CLINICAL TRIAL: NCT06402227
Title: Effectiveness of Board Game on Improving Knowledge, Attitudes and Behavioral Intentions of Infection Control for Senior Elementary School Students: a Randomized Controlled Trial
Brief Title: Effectiveness of Board Game on Improving Elementary School Students' Infection Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HU, HUEY-LAN (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, HU, HUEY-LAN, professor, National Yang Ming Chiao Tung University
Organization: National Yang Ming Chiao Tung University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: NYCU112151AEF
Record Dates: First submitted 2024-04-06; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Knowledge of Infection Control; Attitude of Infection Control; Behavioral Intentions of Infection Control
Keywords: Gamification; Child; Communicable Diseases; Theory of Planned Behavior
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Intervention Model Description: The investigators randomly divided students' classes into the experimental group and the control group. The former received gamified instruction, while the latter received conventional lesson lecture. After a one-month delay, students in the control group were invited to participate in the board game.
Who Masked: Investigator
Masking Description: The Investigator who receives the questionnaires and the Investigator who types the information remain masking.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gamified instruction (Experimental)
  Interventions: Other: gamified instruction
- conventional lesson lecture (Other)
  Interventions: Other: conventional lesson lecture

INTERVENTIONS:
Other: gamified instruction — At the beginning, the speaker played the role of a laboratory rescue team, narrated the background story of the board game, and led the children into the game situation. Then, the speaker explained four types of pathogens, which the investigators defined them according to different types of transmission, including droplets, airborne, blood or body fluids, and fecal-oral. The speaker explained their characteristics and key points, representative diseases in real life, corresponding prevention methods and so on. The lecture lasted for 15 minutes, then the children were divided into different groups to play the board game for about 20 minutes. During the game, students were required to collect "Prevention Method Cards" made by the research team. Students must perform the correct behavior of infection control or answer questions related to the class content in order to obtain the card and win.
  Arms: gamified instruction
Other: conventional lesson lecture — The lecture was about 35 minutes. At the beginning, the speaker explained the terms to children, including infectious diseases, symptoms and pathogens. Next, the speaker introduced the components of the infection chain and how to make infection control behaviors for different parts of it. Then the speaker focused on the four types of transmission, including droplets, airborne, blood or body fluids, and fecal-oral. The speaker illustrated their characteristics and key points, representative diseases in real life, and corresponding prevention methods. In the end, the speaker led the students to practice infection control behaviors, such as the seven correct steps of washing hands, the right steps for wearing and taking off masks, and exercises that can be done to increase immunity.
  Arms: conventional lesson lecture

SUMMARY:
The goal of this clinical trial is to learn if board game can improve elementary school students' infection control intentions. The investigators use the theory of planned behavior (TPB), which includes three main factors: attitude, subjective norm, and perceived behavioral control. The main questions it aims to answer are:

1. Exploring the factors influencing children's behavioral intentions of infection control through theory of planned behavior?
2. The effectiveness of board game on improving children's knowledge and behavioral intentions of infection control?

Researchers will compare gamified instruction to conventional lesson lecture to see if the former has better results.

Students who participated in filled out the questionnaire three times, each time taking about 15 to 20 minutes: before the intervention, after the intervention, and after a one-month delay. The students' legal representatives filled out a basic demographic questionnaire before intervention, which took about 5 minutes.

After a one-month delay, two groups of students were asked to filled out the post-test questionnaire again. Then, students in the control group were invited to participate in a board game and asked which teaching method they preferred (gamified instruction or conventional lesson lecture).

ELIGIBILITY:
Inclusion Criteria:

* Students in fifth to sixth grade of the elementary school (10 to 13 years old) and their legal representatives must fill in the informed consent form.

Exclusion Criteria:

* N/A

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 310 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
intention to infection control behavior | baseline, the day receiving the intervention, a one-month delay after the intervention.
  Theory of planned behavior guided questionnaire (S-CVI/UA=0.962, S-CVI/Ave=0.992) was developed to exam students' attitude, subjective norm, and perceived behavioral control toward infection control behavior over time (pre-intervention, post-intervention, and 4 weeks after intervention). A Likert 5-point scale was used in the TPB questionnaire, the higher the score, the higher the intention for infection control behavior.
knowledge of infection control | baseline, the day receiving the intervention, a one-month delay after the intervention.
  A self-developed knowledge questionnaire (S-CVI/UA=0.8, S-CVI/Ave=0.96) which has fifteen multiple choices questions was used to evaluate students' infection control knowledge over time (pre-intervention, post-intervention, and 4 weeks after intervention). The higher the score, the more positive the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: HUEY-LAN HU, professor, Study Chair — National Yang Ming Chiao Tung University
Locations (1):
- National Yang Ming University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baker RE, Mahmud AS, Miller IF, Rajeev M, Rasambainarivo F, Rice BL, Takahashi S, Tatem AJ, Wagner CE, Wang LF, Wesolowski A, Metcalf CJE. Infectious disease in an era of global change. Nat Rev Microbiol. 2022 Apr;20(4):193-205. doi: 10.1038/s41579-021-00639-z. Epub 2021 Oct 13. PMID 34646006
- [Background] Wang X, Wang S, Wang J, Rong L. A Multiscale Model of COVID-19 Dynamics. Bull Math Biol. 2022 Aug 9;84(9):99. doi: 10.1007/s11538-022-01058-8. PMID 35943625
- [Background] Li DJ, Ko NY, Chang YP, Yen CF, Chen YL. Mediating Effects of Risk Perception on Association between Social Support and Coping with COVID-19: An Online Survey. Int J Environ Res Public Health. 2021 Feb 6;18(4):1550. doi: 10.3390/ijerph18041550. PMID 33561974
- [Background] Cheng HC, Chang YJ, Liao SR, Siewchaisakul P, Chen SL. The impact of COVID-19 on knowledge, attitude, and infection control behaviors among dentists. BMC Oral Health. 2021 Nov 19;21(1):584. doi: 10.1186/s12903-021-01946-w. PMID 34798843
- [Background] Ajzen I. The theory of planned behavior. Organizational Behavior and Human Decision Processes. 1991; 50 (2): 179-211.
- [Background] Luxi N, Giovanazzi A, Capuano A, Crisafulli S, Cutroneo PM, Fantini MP, Ferrajolo C, Moretti U, Poluzzi E, Raschi E, Ravaldi C, Reno C, Tuccori M, Vannacci A, Zanoni G, Trifiro G; Ilmiovaccino COVID19 collaborating group. COVID-19 Vaccination in Pregnancy, Paediatrics, Immunocompromised Patients, and Persons with History of Allergy or Prior SARS-CoV-2 Infection: Overview of Current Recommendations and Pre- and Post-Marketing Evidence for Vaccine Efficacy and Safety. Drug Saf. 2021 Dec;44(12):1247-1269. doi: 10.1007/s40264-021-01131-6. Epub 2021 Nov 5. PMID 34739716
- [Background] Frenck RW Jr, Klein NP, Kitchin N, Gurtman A, Absalon J, Lockhart S, Perez JL, Walter EB, Senders S, Bailey R, Swanson KA, Ma H, Xu X, Koury K, Kalina WV, Cooper D, Jennings T, Brandon DM, Thomas SJ, Tureci O, Tresnan DB, Mather S, Dormitzer PR, Sahin U, Jansen KU, Gruber WC; C4591001 Clinical Trial Group. Safety, Immunogenicity, and Efficacy of the BNT162b2 Covid-19 Vaccine in Adolescents. N Engl J Med. 2021 Jul 15;385(3):239-250. doi: 10.1056/NEJMoa2107456. Epub 2021 May 27. PMID 34043894
- [Background] Wang M, Han X, Fang H, Xu C, Lin X, Xia S, Yu W, He J, Jiang S, Tao H. Impact of Health Education on Knowledge and Behaviors toward Infectious Diseases among Students in Gansu Province, China. Biomed Res Int. 2018 Mar 7;2018:6397340. doi: 10.1155/2018/6397340. eCollection 2018. PMID 29707573
- [Background] Silva MT, Galvao TF, Chapman E, da Silva EN, Barreto JOM. Dissemination interventions to improve healthcare workers' adherence with infection prevention and control guidelines: a systematic review and meta-analysis. Implement Sci. 2021 Oct 24;16(1):92. doi: 10.1186/s13012-021-01164-6. PMID 34689810
- [Background] Alhumaid S, Al Mutair A, Al Alawi Z, Alsuliman M, Ahmed GY, Rabaan AA, Al-Tawfiq JA, Al-Omari A. Knowledge of infection prevention and control among healthcare workers and factors influencing compliance: a systematic review. Antimicrob Resist Infect Control. 2021 Jun 3;10(1):86. doi: 10.1186/s13756-021-00957-0. PMID 34082822
- [Background] McCoy L, Lewis JH, Dalton D. Gamification and Multimedia for Medical Education: A Landscape Review. J Am Osteopath Assoc. 2016 Jan;116(1):22-34. doi: 10.7556/jaoa.2016.003. PMID 26745561
- [Background] Sardi L, Idri A, Fernandez-Aleman JL. A systematic review of gamification in e-Health. J Biomed Inform. 2017 Jul;71:31-48. doi: 10.1016/j.jbi.2017.05.011. Epub 2017 May 20. PMID 28536062
- [Background] Guan X, Sun C, Hwang G, Xue K, Wang Z. Applying game-based learning in primary education: a systematic review of journal publications from 2010 to 2020. Interactive Learning Environments. 2022; null 1-23.
- [Background] de Graaf M, Beck R, Caccio SM, Duim B, Fraaij P, Le Guyader FS, Lecuit M, Le Pendu J, de Wit E, Schultsz C. Sustained fecal-oral human-to-human transmission following a zoonotic event. Curr Opin Virol. 2017 Feb;22:1-6. doi: 10.1016/j.coviro.2016.11.001. Epub 2016 Nov 23. PMID 27888698
- [Background] Wolfe ND, Dunavan CP, Diamond J. Origins of major human infectious diseases. Nature. 2007 May 17;447(7142):279-83. doi: 10.1038/nature05775. PMID 17507975
- [Background] Viana Martins CP, Xavier CSF, Cobrado L. Disinfection methods against SARS-CoV-2: a systematic review. J Hosp Infect. 2022 Jan;119:84-117. doi: 10.1016/j.jhin.2021.07.014. Epub 2021 Oct 18. PMID 34673114
- [Background] Heijne JC, Teunis P, Morroy G, Wijkmans C, Oostveen S, Duizer E, Kretzschmar M, Wallinga J. Enhanced hygiene measures and norovirus transmission during an outbreak. Emerg Infect Dis. 2009 Jan;15(1):24-30. doi: 10.3201/eid1501.080299. PMID 19116045
- [Background] Baden LR, El Sahly HM, Essink B, Kotloff K, Frey S, Novak R, Diemert D, Spector SA, Rouphael N, Creech CB, McGettigan J, Khetan S, Segall N, Solis J, Brosz A, Fierro C, Schwartz H, Neuzil K, Corey L, Gilbert P, Janes H, Follmann D, Marovich M, Mascola J, Polakowski L, Ledgerwood J, Graham BS, Bennett H, Pajon R, Knightly C, Leav B, Deng W, Zhou H, Han S, Ivarsson M, Miller J, Zaks T; COVE Study Group. Efficacy and Safety of the mRNA-1273 SARS-CoV-2 Vaccine. N Engl J Med. 2021 Feb 4;384(5):403-416. doi: 10.1056/NEJMoa2035389. Epub 2020 Dec 30. PMID 33378609
- [Background] Nieman DC, Sakaguchi CA. Physical activity lowers the risk for acute respiratory infections: Time for recognition. J Sport Health Sci. 2022 Nov;11(6):648-655. doi: 10.1016/j.jshs.2022.08.002. Epub 2022 Aug 20. PMID 35995362
- [Background] Iddir M, Brito A, Dingeo G, Fernandez Del Campo SS, Samouda H, La Frano MR, Bohn T. Strengthening the Immune System and Reducing Inflammation and Oxidative Stress through Diet and Nutrition: Considerations during the COVID-19 Crisis. Nutrients. 2020 May 27;12(6):1562. doi: 10.3390/nu12061562. PMID 32471251
- [Background] Mercola J, Grant WB, Wagner CL. Evidence Regarding Vitamin D and Risk of COVID-19 and Its Severity. Nutrients. 2020 Oct 31;12(11):3361. doi: 10.3390/nu12113361. PMID 33142828
- [Background] Talic S, Shah S, Wild H, Gasevic D, Maharaj A, Ademi Z, Li X, Xu W, Mesa-Eguiagaray I, Rostron J, Theodoratou E, Zhang X, Motee A, Liew D, Ilic D. Effectiveness of public health measures in reducing the incidence of covid-19, SARS-CoV-2 transmission, and covid-19 mortality: systematic review and meta-analysis. BMJ. 2021 Nov 17;375:e068302. doi: 10.1136/bmj-2021-068302. PMID 34789505
- [Background] White KM, Jimmieson NL, Obst PL, Graves N, Barnett A, Cockshaw W, Gee P, Haneman L, Page K, Campbell M, Martin E, Paterson D. Using a theory of planned behaviour framework to explore hand hygiene beliefs at the '5 critical moments' among Australian hospital-based nurses. BMC Health Serv Res. 2015 Feb 13;15:59. doi: 10.1186/s12913-015-0718-2. PMID 25888894
- [Background] Shubayr MA, Mashyakhy M, Al Agili DE, Albar N, Quadri MF. Factors Associated with Infection-Control Behavior of Dental Health-Care Workers During the COVID-19 Pandemic: A Cross-Sectional Study Applying the Theory of Planned Behavior. J Multidiscip Healthc. 2020 Nov 12;13:1527-1535. doi: 10.2147/JMDH.S278078. eCollection 2020. PMID 33209032
- [Background] Cox JL, Simpson MD, Letts WJ, Cavanagh HM. A. Re-thinking microbiology/infection control education to enhance the practice-readiness of health professional students: More than just a curriculum issue. Journal of Learning Design. 2015; 8 (1): 55-67.
- [Background] Zomordi G, Moradi M, Hasanzadeh M, Ghavami V. The effect of education based on the theory of planned behavior on the intention of vaccination against human papillomavirus in female students: A controlled educational trial. J Educ Health Promot. 2022 Jul 29;11:237. doi: 10.4103/jehp.jehp_1145_21. eCollection 2022. PMID 36177425
- [Background] van Gaalen AEJ, Brouwer J, Schonrock-Adema J, Bouwkamp-Timmer T, Jaarsma ADC, Georgiadis JR. Gamification of health professions education: a systematic review. Adv Health Sci Educ Theory Pract. 2021 May;26(2):683-711. doi: 10.1007/s10459-020-10000-3. Epub 2020 Oct 31. PMID 33128662
- [Background] Hale AR, Young VL, Grand A, McNulty CA. Can Gaming Increase Antibiotic Awareness in Children? A Mixed-Methods Approach. JMIR Serious Games. 2017 Mar 24;5(1):e5. doi: 10.2196/games.6420. PMID 28341618
- [Background] Banos RM, Cebolla A, Oliver E, Alcaniz M, Botella C. Efficacy and acceptability of an Internet platform to improve the learning of nutritional knowledge in children: the ETIOBE Mates. Health Educ Res. 2013 Apr;28(2):234-48. doi: 10.1093/her/cys044. Epub 2012 Apr 11. PMID 22498924
- [Background] Lakshman RR, Sharp SJ, Ong KK, Forouhi NG. A novel school-based intervention to improve nutrition knowledge in children: cluster randomised controlled trial. BMC Public Health. 2010 Mar 10;10:123. doi: 10.1186/1471-2458-10-123. PMID 20219104
- [Background] Suleiman-Martos N, Garcia-Lara RA, Martos-Cabrera MB, Albendin-Garcia L, Romero-Bejar JL, Canadas-De la Fuente GA, Gomez-Urquiza JL. Gamification for the Improvement of Diet, Nutritional Habits, and Body Composition in Children and Adolescents: A Systematic Review and Meta-Analysis. Nutrients. 2021 Jul 20;13(7):2478. doi: 10.3390/nu13072478. PMID 34371989
- See also: Introduction to the chain of infection — https://archive.cdc.gov/www_cdc_gov/csels/dsepd/ss1978/lesson1/section10.html
- See also: Introduction to the Theory of Planed Behavior — https://epaper.naer.edu.tw/edm.php?grp_no=2&edm_no=51&content_no=1421